CLINICAL TRIAL: NCT02050893
Title: The Effect of Midazolam on Fluid Responsiveness in Septic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Department of critical care medicine, Zhongda Hospital, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fluid responsiveness
Record Dates: First submitted 2013-03-05; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Septic Shock
Keywords: septic shock; sepsis; fluid responsiveness; Midazolam; Propofol; haemodynamics
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam (Experimental): Midazolam infused at a 0.03mg/kg loading dose ,and 0.02-0.1mg/kg.h maintenance dose to achieve Ramsay score of 4
  Interventions: Drug: sedatives(Midazolam and Propofol)
- Propofol (Experimental): Propofol infuse at a loading dose of 0.5mg/kg，and 0.5-2.0mg/kg.h maintenance dose to achieve Ramsay score of 4
  Interventions: Drug: sedatives(Midazolam and Propofol)

INTERVENTIONS:
Drug: sedatives(Midazolam and Propofol)

SUMMARY:
Fluid resuscitation remains the foundation for septic treatment.The evaluation of fluid responsiveness has significance in volume resuscitation for septic shock patients. As the sedative which is commonly used in ICU, Midazolam is supposed to change fluid responsiveness for the pharmacological effect of venodilation. However, the hypothesis has not been certified clinically. In this research, the investigators aim to test the hypothesis that Midazolam can increase fluid responsiveness(using passive leg raising test) in septic shock patients.

ELIGIBILITY:
Patients are included if they meet the following inclusion criteria:

1. Above 18 years old
2. Endotracheal intubated and mechanical ventilated
3. Awake, can communicate with researchers
4. Diagnosed as septic shock. The definition of septic shock was clarified in Year 2001 ACCP/SCCM guidelines
5. Within 24 hours after the EGDT resuscitation goals are achieved
6. Informed consent are signed.

Exclusion Criteria

1. Under 18 years old
2. Intra-abdominal hypertension
3. Central nerves system dysfunction
4. Heart failure and other cardiac dysfunction such as cardiac conduction block,acute coronary syndrome, cardiogenic shock
5. Proof of volume overload or contradiction of fluid infusion
6. Existence of arterial aneurysm, serious valvular disease,extensive peripheral vascular occlusion disease and insertion of artificial pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
percentage of participants with more than 10% increase of cardiac index by passive leg raising after sedation | Baseline,after sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care , Zhong-da Hospital, Nanjing, Jiangsu, China